CLINICAL TRIAL: NCT06879600
Title: Research on Pre-Anesthetic Blood Oxygenation Effect of High-Flow Nasal Oxygen for Emergency Surgery Patients With Full Stomachs
Brief Title: High-Flow Nasal Oxygen for Preoxygenation in Emergency Surgery Patients With Full Stomachs
Acronym: HFNC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nguyen Dang Thu (Other)
Collaborators: Hanoi Medical University (Other); Phu Tho General Hospital (Unknown)
Responsible Party: Sponsor-Investigator, Nguyen Dang Thu, Ph.D; M.D., Vietnam Military Medical University
Organization: Vietnam Military Medical University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HongGMHS-No.1185; NCS42HFNC (Other: Hanoi Medical University)
Record Dates: First submitted 2025-03-05; First posted 2025-03-17 (Actual); Last update posted 2025-03-17 (Actual); Status verified 2025-03

CONDITIONS: High-flow Nasal Cannula; Oxygenation; General Anesthesia; Induction Anesthesia; Emergency Surgery Patients; Full Stomach
Keywords: High-flow nasal cannula; oxygenation; Induction anesthesia; Emergency Surgery Patients; full stomach

STUDY DESIGN:
Intervention Model Description: prospective, single-center, randomized controlled trial
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High-flow nasal cannula therapy application (Active Comparator): Intervention Group: Patients will undergo HFNC preoxygenation for 3 minutes with a flow rate of 60 L/min of heated and humidified pure oxygen (100% FiO₂, 37°C - Optiflow; Fisher & Paykel Healthcare, Auckland, New Zealand). To minimize air contamination, large or medium nasal cannulae will be selected based on the patient's nostril size. During the intubation process, HFNC will be maintained to facilitate either:
  Continuous oxygenation while the patient breathes spontaneously, or Apneic oxygenation during laryngoscopy for rapid sequence intubation (RSI).
  Interventions: Device: High-flow nasal cannula therapy application
- Traditional facemask (Placebo Comparator): Control Group: Patients will undergo preoxygenation for 3 minutes using a face mask (sized appropriately to fit the patient and ensure an airtight seal) connected to an Aisys CS2 ventilation system (General Electric, GE Healthcare, Oy, Finland). In this group, the ventilation system will be set with a fresh gas flow of 10 L/min, FiO₂ = 100%, without inspiratory support or expiratory positive pressure. The face mask (Economy, Intersurgical, Fontenay-sous-Bois, France) will be removed after induction to enable intubation.
  Interventions: Device: Traditional facemask

INTERVENTIONS:
Device: High-flow nasal cannula therapy application — Patients will undergo HFNC preoxygenation for 3 minutes with a flow rate of 60 L/min of heated and humidified pure oxygen (100% FiO₂, 37°C - Optiflow; Fisher & Paykel Healthcare, Auckland, New Zealand). To minimize air contamination, large or medium nasal cannulae will be selected based on the patient's nostril size
  Arms: High-flow nasal cannula therapy application
Device: Traditional facemask — Patients will undergo preoxygenation for 3 minutes using a face mask (sized appropriately to fit the patient and ensure an airtight seal) connected to an Aisys CS2 ventilation system (General Electric, GE Healthcare, Oy, Finland). In this group, the ventilation system will be set with a fresh gas flow of 10 L/min, FiO₂ = 100%, without inspiratory support or expiratory positive pressure. The face mask (Economy, Intersurgical, Fontenay-sous-Bois, France) will be removed after induction to enable intubation.
  Arms: Traditional facemask

SUMMARY:
Patients with full stomachs face a high risk of regurgitation and aspiration under general anesthesia. To minimize the time between the loss of airway protective reflexes and successful tracheal intubation, rapid sequence induction intubation is commonly used. However, these patients are particularly vulnerable to hypoxemia during anesthesia induction, especially in emergency cases. Pre-oxygenation before induction is crucial for ensuring patient safety during apnea.

High-flow nasal oxygen (HFNO) therapy, which consists of an air/oxygen blender, an active humidifier, and a single heated circuit, has recently gained widespread use in intensive care units (ICUs) for managing hypoxemic respiratory failure. HFNC can deliver a constant fraction of inspired oxygen (FiO₂) from 0.21 to 1.0 at high flow rates (up to 60 L/min or higher). Its advantages include generating continuous positive airway pressure, reducing anatomical dead space, improving ventilation-perfusion matching, enhancing mucociliary clearance, and decreasing the work of breathing.

Given these benefits, HFNO has the potential to improve pre-oxygenation before and during anesthesia induction in emergency surgery patients with full stomachs.

DETAILED DESCRIPTION:
This is a prospective, single-center, randomized controlled trial designed to evaluate the effects of HFNO on preoxygenation before and during anesthesia induction in emergency surgery patients with full stomachs. Adult patients undergoing emergency surgery with general anesthesia will be enrolled in the study.

After obtaining written informed consent, patients will be randomly assigned to one of the study groups:

- Intervention Group: Patients will undergo HFNO preoxygenation for 3 minutes with a flow rate of 60 L/min of heated and humidified pure oxygen (100% FiO₂, 37°C - Optiflow; Fisher & Paykel Healthcare, Auckland, New Zealand). To minimize air contamination, large or medium nasal cannulae will be selected based on the patient's nostril size. During the intubation process, HFNO will be maintained to facilitate either: Continuous oxygenation while the patient breathes spontaneously, or Apneic oxygenation during laryngoscopy for rapid sequence intubation (RSI).

- Control Group: Patients will undergo preoxygenation for 3 minutes using a face mask (sized appropriately to fit the patient and ensure an airtight seal) connected to an Aisys CS2 ventilation system (General Electric, GE Healthcare, Oy, Finland). In this group, the ventilation system will be set with a fresh gas flow of 10 L/min, FiO₂ = 100%, without inspiratory support or expiratory positive pressure. The face mask (Economy, Intersurgical, Fontenay-sous-Bois, France) will be removed after induction to enable intubation.

Rapid sequence induction and intubation were performed using fentanyl (2 mcg/kg), propofol (2 mg/kg), and rocuronium (1 mg/kg). Intubation was performed 90 seconds after rocuronium administration. Cricoid pressure was applied from the moment the patient lost consciousness until intubation was successfully completed.

The current guidelines advise interrupting intubation to focus on oxygenation (ie, face mask ventilation) for oxygen desaturation ≤94%.

ELIGIBILITY:
Inclusion Criteria:

* Emergency surgical patients at risk of gastric fullness requiring endotracheal intubation.
* Patients aged 18 years or older.
* Health status classified as ASA I or II.
* Mallampati classification I or II.

Exclusion Criteria:

* Patients with a predicted difficult airway, facial deformities, or an inability to achieve a proper mask seal.
* Patients with respiratory diseases.
* Pregnant patients.
* Patients allergic to anesthesia or resuscitation drugs.
* Patients who do not consent to participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2023-07-19 (Actual); Primary Completion 2026-12-15 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
PaO2 | Perioperative
  PaO2 was checked via arterial blood gas at different time points
Changes SpO2 during 3 minutes of preoxygenation | Perioperative
  SpO2 was recorded at baseline (before preoxygenation) and every 30 seconds during 3 minutes of preoxygenation
Incidence of desaturation during rapid sequence induction anesthesia | Periprocedural
  Desaturation is defined as SpO2 < 94% during apnea and intubation period of induction anesthesia
Number of episode of facemask ventilation during apnea period | Periprocedural
  during apnea period, if SpO2 < 94% facemask ventilation will be applied

SECONDARY OUTCOMES:
Changes TcCO2 | Periprocedural
  Continuous transcutaneous CO2 partial pressure monitoring (TcCO2). TcCO2 was monitored with a sensor (V-Sign™ 2 sensor; SenTec, Switzerland) attached to the skin of the forearm or anterior chest, connected to the SenTec digital display after calibration. TcCO2 was recorded every 30 seconds during preoxygenation, apnea and intubation period
Gastric volume | Perioperative
  Gastric volume assessment was accessed using ultrasound
Incidence of regurgitation and aspiration | Periprocedural
  regurgitation and aspiration were checked during laryngoscopy
Nasal congestion | 1 hour after extubation
  Evaluate after extubation
Hemodynamic effects | During 3 minutes of preoxygenation
  Any events of bradycardia, tachycardia, hypertension, or hypotension during preoxygenation period were recorded

CONTACTS AND LOCATIONS:
Overall Officials: Lam Nguyen Duc, Assoc.Prof, PhD, MD, Study Director — Hanoi Medical University
Locations (1):
- Department of Anesthesia, Phu Tho General Hospital, Việt Trì, Phu Tho, Vietnam

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Vargas F, Saint-Leger M, Boyer A, Bui NH, Hilbert G. Physiologic Effects of High-Flow Nasal Cannula Oxygen in Critical Care Subjects. Respir Care. 2015 Oct;60(10):1369-76. doi: 10.4187/respcare.03814. Epub 2015 May 5. PMID 25944940
- [Background] Vourc'h M, Asfar P, Volteau C, Bachoumas K, Clavieras N, Egreteau PY, Asehnoune K, Mercat A, Reignier J, Jaber S, Prat G, Roquilly A, Brule N, Villers D, Bretonniere C, Guitton C. High-flow nasal cannula oxygen during endotracheal intubation in hypoxemic patients: a randomized controlled clinical trial. Intensive Care Med. 2015 Sep;41(9):1538-48. doi: 10.1007/s00134-015-3796-z. Epub 2015 Apr 14. PMID 25869405
- [Background] Patel A, Nouraei SA. Transnasal Humidified Rapid-Insufflation Ventilatory Exchange (THRIVE): a physiological method of increasing apnoea time in patients with difficult airways. Anaesthesia. 2015 Mar;70(3):323-9. doi: 10.1111/anae.12923. Epub 2014 Nov 10. PMID 25388828
- [Background] Badiger S, John M, Fearnley RA, Ahmad I. Optimizing oxygenation and intubation conditions during awake fibre-optic intubation using a high-flow nasal oxygen-delivery system. Br J Anaesth. 2015 Oct;115(4):629-32. doi: 10.1093/bja/aev262. Epub 2015 Aug 7. PMID 26253608
- [Background] Lodenius A, Piehl J, Ostlund A, Ullman J, Jonsson Fagerlund M. Transnasal humidified rapid-insufflation ventilatory exchange (THRIVE) vs. facemask breathing pre-oxygenation for rapid sequence induction in adults: a prospective randomised non-blinded clinical trial. Anaesthesia. 2018 May;73(5):564-571. doi: 10.1111/anae.14215. Epub 2018 Jan 13. PMID 29330853
- [Derived] Lam ND, Son LDT, Phat TM, Thu ND, Nga NT, Son VT, Hong BM. High-flow nasal oxygen versus face-mask ventilation for rapid sequence induction in non-elective surgical patients: a randomized controlled trial. BMC Anesthesiol. 2026 Jan 31. doi: 10.1186/s12871-026-03654-w. Online ahead of print. PMID 41620676